CLINICAL TRIAL: NCT03510286
Title: Validation of a Protein Creatinine (PrCr) Dipstick Diagnostic Test for Proteinuria Screening in Antenatal Care Clinics in Ghana
Brief Title: Validation of a PrCr Dipstick Diagnostic Test in Ghana
Status: Completed | Type: Observational
Sponsor: PATH (Other)
Collaborators: Kintampo Health Research Centre, Ghana (Other); United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 1133673-2
Record Dates: First submitted 2018-04-17; First posted 2018-04-27 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2019-08

CONDITIONS: Proteinuria; Preeclampsia
Keywords: proteinuria; preeclampsia; diagnostic; dipstick; protein; urine; creatinine
MeSH Terms: conditions — Proteinuria; Pre-Eclampsia; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Pregnant women: Pregnant women attending ANC clinics in Techiman Holy Family Hospital and Kintampo North and South districts (all hospitals and clinics inclusive where ANC services are provided) are the primary participant group- primarily women of reproductive age. Pregnant women attending routine ANC will be enrolled. In addition to routine ANC, pregnant women will be tested with the Test-it™ PrCr Urinalysis Strips. Pregnant women are a potentially vulnerable population whose participation in this research is necessary given the target use case for this diagnostic tool: providing reliable and accurate point of care screening of proteinuria in ANC settings. The legal age of consent in Ghana is 18 years and women under the age of 18 will not be recruited for this study.
  Interventions: Diagnostic Test: Test-it™ PrCr Urinalysis Strips

INTERVENTIONS:
Diagnostic Test: Test-it™ PrCr Urinalysis Strips — The LifeAssay Diagnostics prototype PrCr dipstick has been designed to provide the measurement of both protein and creatinine while retaining a very low estimated cost that is comparable to the current protein-only dipsticks at $0.06-0.10 per test. In 2015, an initial laboratory-based validation study of the prototype LAD PrCr test was used on more than 500 characterized urine samples from pregnant women. This validation study demonstrated comparable accuracy for detection of severe proteinuria of the LAD PrCr test to the much more expensive commercial POC test available for PrCr determination, the Siemens Multistix® PRO 10LS. These results were compared to laboratory-based reference standard assays for proteinuria measurement.

SUMMARY:
This evaluation will aim to generate a body of evidence that will determine performance characteristics of the current PrCr dipstick test and the feasibility of its use in target ANC settings. Data will be used to inform further product development and/or support development of an introduction framework, including the process and associated resources needed for incorporation of the PrCr test into future larger-scale demonstration studies as well as to support early product launch.

The objectives of the evaluation are as follows:

Primary objective: Assess the accuracy of the PrCr dipstick test for detection of proteinuria in representative antenatal care settings in Ghana.

Exploratory objectives:

* Understand the feasibility of integrating the use of the PrCr test into ANC services in Ghana.
* Explore the potential for improved ANC management of PE/E using the PrCr test in intended ANC settings versus the current standard of care used for proteinuria screening, protein-only determination via a low -cost urine dipstick test.

DETAILED DESCRIPTION:
This cross-sectional diagnostic accuracy evaluation will employ mixed methods to assess the performance of the PrCr dipstick test and to explore the operational feasibility of using this test as an alternative to the current protein-only test. These methods include:

Assess the accuracy of the PrCr test for detection of proteinuria in a representative ANC setting in Ghana.

• Detection of proteinuria using the PrCr dipstick test compared to the current standard of care and laboratory reference assay used for confirming proteinuria. Patient samples will be tested with multiple assays. The PrCr test and a protein-only dipstick (The Mission® Urinalysis Reagent Strips (Urine), will be used at the point of care. Patient samples will be transferred to KHRC laboratory using cold boxes (conditioned at 2oC - 8oC) and will be tested using a laboratory reference assay.

Understand the feasibility of integrating the use of the PrCr test into ANC services.

* Pre- and post-evaluation of ANC staff training on use of the PrCr test
* Interviews with ANC staff
* Consultations with key district and national stakeholders.

Explore the potential for improved ANC management of PE/E using the PrCr test in the intended ANC setting.

* Analysis of pregnancy outcomes (live or stillbirth) and review of referral records. Actual outcomes along with referral practices and linkage to care based on the current diagnostics will be compared to any potential changes in referral practices and linkage to care based on prospective PrCr test results.
* Assessment of use of PrCr test with other clinical indicators and integration into diagnostic algorithms. Prospective PrCr test results will be integrated into an existing diagnostic algorithm to assess any potential changes in referral practices and linkage to care.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman 18 years of age or older (self-report)
* Attending a study site facility for ANC
* ANC visit is within the final 12 weeks of pregnancy (within 12 weeks or less before expected due date)
* Willing to provide written informed consent for study participation

Exclusion Criteria:

* ANC visit is not within the final 12 weeks of pregnancy
* Unwilling to provide written informed consent for study participation
* Pregnant woman less than 18 years of age

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women
Study Population: Pregnant women attending ANC clinics in Techiman Holy Family Hospital and Kintampo North and South districts (all hospitals and clinics inclusive where ANC services are provided) are the primary participant group- primarily women of reproductive age. Pregnant women are a potentially vulnerable population whose participation in this research is necessary given the target use case for this diagnostic tool: providing reliable and accurate point of care screening of proteinuria in ANC settings. The legal age of consent in Ghana is 18 years and women under the age of 18 will not be recruited for this study.
Sampling Method: Non-Probability Sample
Enrollment: 1483 (Actual)
Dates: Start 2018-09-30 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Accuracy of the PrCr dipstick test compared to a laboratory reference assay (chemistry analyzer measurement of protein and creatinine) | September 20198-February 2019
  The results of the PrCr dipstick test will be compared to the results of a laboratory reference assay. Sensitivity and specificity analyses will be conducted at thresholds for normal and proteinuria.
Accuracy of the PrCr dipstick test compared to a protein only dipstick. | September 20198-February 2019
  The results of the PrCr dipstick test will be compared to the results of the protein only test. Sensitivity and specificity analyses will be conducted at thresholds for normal and proteinuria.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Newton, PhD, Principal Investigator — Kintampo Health Research Centre, Ghana
Locations (1):
- Kintampo Health Research Center, Kintampo, Ghana

IPD SHARING:
Plan to Share IPD: No